CLINICAL TRIAL: NCT06654544
Title: Prevalence and Clinical Features of Intracerebral Hemorrhage Among Stroke Patients Admitted to Assiut University Hospital
Brief Title: Epidemiology of Intracerebral Hemorrhage
Acronym: ICH
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Norhan Mohamed Hassan Bakri, Principal Investigator, Assiut University
Other Study IDs: 200913
Record Dates: First submitted 2024-10-14; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: ICH - Intracerebral Hemorrhage
Keywords: prevalence; ich
MeSH Terms: conditions — Cerebral Hemorrhage; Hepatitis, Infectious Canine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Exploring the risk factors and associations of intracerebral hemorrhage

DETAILED DESCRIPTION:
Exploring the clinical characteristics and prevalence of intracerebral hemorrhage in Assiut University

ELIGIBILITY:
Inclusion Criteria:

* both sex
* Age ≥ 18
* patients diagnosed with non traumatic hemorrhagic stroke on brain computed tomography scan

Exclusion Criteria:

* presence of space occupying lesion visible on brain computed tomography scan
* preceding brain trauma or post traumatic cerebral hemorrhagic stroke
* presence of ischemic stroke
* presence hemorrhagic transformation on top of acute ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke Patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Volume of Intracerebral Hemorrhage Among Stroke Patients Admitted to Assiut University Hospital | At time of enrollment of study and after 24 hours
  CT data (ABC/2) formula for intracerebral hemorrhage volume

CONTACTS AND LOCATIONS:
Overall Officials: Norhan MH Bakri, MD, Principal Investigator — Assiut University; Ahmed NasrEldein, Ass.Professor, Study Director — Assiut University

REFERENCES:
- [Result] An SJ, Kim TJ, Yoon BW. Epidemiology, Risk Factors, and Clinical Features of Intracerebral Hemorrhage: An Update. J Stroke. 2017 Jan;19(1):3-10. doi: 10.5853/jos.2016.00864. Epub 2017 Jan 31. PMID 28178408